CLINICAL TRIAL: NCT03680716
Title: Analgesic Efficacy of a Combined Saphenous Nerve Block and IPACK Block Versus Local Infiltration Analgesia After Anterior Cruciate Ligament Reconstruction: a Randomized Controlled Double-blinded Trial.
Brief Title: Combined Saphenous Nerve and IPACK Blocks Versus Infiltration Analgesia After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program director of regional anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER 2018-01163
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Anterior Cruciate Ligament Injury; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Pain, Postoperative; Anterior Cruciate Ligament Injuries | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPACK block (Experimental): Saphenous nerve block and IPACK block by anesthetist under ultrasound guidance.
  Interventions: Drug: Ropivacaine injection
- Local infiltration analgesia (Active Comparator): Periarticular infiltration by surgeon
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — Saphenous nerve block with 20ml of ropivacaine 0.5% and IPACK block with 30ml of ropivacaine 0.2% (total dose of 160 mg).
  Arms: IPACK block
Drug: Ropivacaine injection — Periarticular infiltration of 80 ml ropivacaine 0.2% (total dose of 160mg).
  Arms: Local infiltration analgesia

SUMMARY:
A lot of patient have posterior knee pain after ACL reconstruction despite saphenous nerve block. Recently a new block has been described, know as IPACK block (interspace between the popliteal artery and the capsule of the posterior knee). The objective of this randomized controlled double-blinded trial is to assess whether a combined saphenous nerve block with IPACK block is more effective for the postoperative pain than a local infiltration analgesia.

DETAILED DESCRIPTION:
The saphenous nerve and the iPACK will be performed after general anaesthesia induction and before the surgery under ultrasound-guidance.

The local infiltration analgesia will be performed by the surgeon during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Statut ASA I-III.
* Patient scheduled for anterior crutiate ligament reconstruction under general anesthesia.

Exclusion Criteria:

* Pregnancy.
* Contraindication to local anesthesia.
* Patient with chronic pain, opioid consumption or alcohol consumption.
* Patient with coagulation trouble, hepatic dysfunction or renal dysfunction.
* Patient with diabetic or femoral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption (mg) | 24 hours postoperatively

SECONDARY OUTCOMES:
Total morphine consumption (mg) | 2 hours, 48 hours and 72 hours postoperatively
Pain scores (numeric rating scale, 0-10) at rest and on movement | 2hours, 24hours, 48hours and 72hours postoperatively
  0= no pain, 10=the worst pain imaginable
Rate of postoperative nausea and vomiting | 2hours, 24hours, 48hours and 72hours postoperatively
  Yes/No
Rate of antiemetic consumption | 2hours, 24hours, 48hours and 72hours postoperatively
  Yes/No
Rate of pruritus | 2hours, 24hours, 48hours and 72hours postoperatively
  Yes/No
Active flexion | 24hours, 48hours and 72hours postoperatively
  Flexion of the knee by the patient measured in degrees
Quadriceps muscle strength (numeric scale, 1-5) | 24hours, 48hours and 72hours postoperatively
  1=no contraction, 5=normal strength
Distance walked (meters) | 24 hours, 48hours and 72hours postoperatively
Anterior Cruciate Ligament - Return to Sport after Injury survey | 4 and 8 postoperative months
International Knee Documentation Committee score | 4 and 8 postoperative months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martin R, Kirkham KR, Ngo THN, Gonvers E, Lambert J, Albrecht E. Combination of femoral triangle block and infiltration between the popliteal artery and the capsule of the posterior knee (iPACK) versus local infiltration analgesia for analgesia after anterior cruciate ligament reconstruction: a randomized controlled triple-blinded trial. Reg Anesth Pain Med. 2021 Sep;46(9):763-768. doi: 10.1136/rapm-2021-102631. Epub 2021 May 26. PMID 34039734